CLINICAL TRIAL: NCT00103636
Title: Peripheral Venous Catheter Trial: 3 Day Versus No Routine Change
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Brisbane and Women's Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBWH 2003/131
Record Dates: First submitted 2005-02-11; First posted 2005-02-14 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-02

CONDITIONS: Phlebitis
Keywords: Phlebitis/etiology; Infusions; Intravenous/adverse effects; Randomised controlled trial; Phlebitis/prevention; Adult; Time factors
MeSH Terms: conditions — Phlebitis

INTERVENTIONS:
Procedure: Extending peripheral intravenous (IV) cannula dwell times

SUMMARY:
The purpose of this study is to investigate the effects of extending the dwell time of peripheral intravenous cannulas on clinical outcomes and cost.

DETAILED DESCRIPTION:
Among hospitalized patients, intravenous therapy is the most common invasive procedure. It is associated with a phlebitis rate of between 1.1% and 63% and a central venous catheter related bacteremia rate of approximately 3.0%. Catheter related blood-stream infections have an attributable mortality rate of 12% to 25%. Factors thought to be associated with these complications include insertion techniques, catheter securement, type of catheter used, type of infusate and additives, post-insertion catheter care and length of time the catheter remains in place.

Current Centers of Disease Control Guidelines provide direction for intravenous therapy management including a recommendation that peripheral intravenous catheters should be re-sited every 72-96 hours. Data underpinning the recommendation was collected in 1992, over a decade ago. Since that time, there have been improvements in catheter design and composition, and prospective surveillance studies have demonstrated the safety of longer dwell times. To date, these observations have not been validated in adults, using randomized controlled trial methodology.

Re-siting intravenous cannulas causes discomfort to patients and has a high recurrent cost. The primary aim of the present study is to compare the rates of peripheral catheter-related blood stream infection, catheter-related local infection, phlebitis and obstruction between two groups of patients - those having routine catheter changes every 72 hours and those having catheter changes only when clinically indicated.

Specific hypotheses:

That changing intravenous peripheral catheters when indicated by clinical signs compared to changing intravenous catheters every 3 days reduces the incidence of intravenous catheter related morbidity.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to join the Peripheral Venous Catheter Trial if:

* They are inpatients at the Royal Brisbane and Royal Women's Hospital who are at least 18 years of age

AND

* They are scheduled or expected to have a peripheral venous catheter indwelling for at least 4 days.

AND

* They have had their catheter inserted by a nurse from the IV Therapy Team

Exclusion Criteria:

* Patients with an existing bloodstream infection
* Those receiving immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-03; Study Completion 2004-12

PRIMARY OUTCOMES:
Phlebitis during the course of the infusion and up to 48 hours after peripheral venous catheter removal

SECONDARY OUTCOMES:
Infiltration permeation of IV fluid into the interstitial compartment
Local infection at the site of the catheter
Catheter-related blood stream infection
Catheter colonization
Cost

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia